CLINICAL TRIAL: NCT00869934
Title: Cognitive-Behavior Therapy for Insomnia: Component Analysis and Treatment
Brief Title: Cognitive-Behavior Therapy for Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Charles M. Morin, Professeur, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH079188-02 (NIH); NIMH
Record Dates: First submitted 2009-03-24; First posted 2009-03-26 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Insomnia
Keywords: Insomnia; Sleep disorders; Treatment; Sleep disturbances
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Parasomnias | interventions — Cognitive Behavioral Therapy; Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1. Cognitive-Behavior Therapy (Active Comparator)
  Interventions: Other: Cognitive-Behavior Therapy
- 2. Behavior Therapy (Experimental)
  Interventions: Other: Behavior Therapy
- 3. Cognitive Therapy (Experimental)
  Interventions: Other: Cognitive Therapy

INTERVENTIONS:
Other: Cognitive-Behavior Therapy — Sleep restriction, stimulus control, cognitive therapy
  Arms: 1. Cognitive-Behavior Therapy
Other: Behavior Therapy — Sleep restriction and stimulus control
  Arms: 2. Behavior Therapy
Other: Cognitive Therapy — Cognitive restructuring therapy
  Arms: 3. Cognitive Therapy

SUMMARY:
Insomnia is a prevalent public health problem affecting large segments of the population on an occasional, recurrent, or chronic basis. Persistent insomnia is associated with impairments in daytime functioning, reduced quality of life, and increased health-care costs. Despite evidence that cognitive-behavior therapy (CBT) is an effective and well accepted treatment for insomnia, a significant proportion of individuals do not respond adequately to this treatment. Hence, there is a need to identify the active therapy components and mechanisms of change in order to develop more effective therapeutic approaches and optimize outcomes. The specific aims of the proposed study are to (a) evaluate the effects of behavioral versus cognitive therapies for insomnia and associated daytime impairment, (b) investigate the mechanisms of change and, (c) examine the impact of insomnia therapies on psychiatric conditions commonly associated with insomnia (anxiety disorders and depression). A sample of 186 adults with chronic insomnia will be recruited from two sites (Laval University and University of California, Berkeley). Participants will be randomly assigned to one of three groups: (a) behavior therapy (BT; n = 62), (b) cognitive therapy (CT; n = 62), or (c) cognitive-behavior therapy (CBT; n = 62). Measures of outcome (sleep/insomnia, daytime functioning) will be administered at baseline, end of treatment, and at 6- and 12-month follow up. Measures of mechanisms of change (maladaptive sleep habits, unhelpful beliefs, sleep-related worry) will be administered at baseline, after the 4th and 8th therapy sessions, and at the end of treatment. It is expected that (1) BT and CBT will be more effective for improving sleep, relative to CT, (2) CT and CBT will be more effective for reducing daytime functional impairment, relative to BT and (3)CT will be more effective than BT in reducing comorbid psychiatric disorders. The public health significance of the proposed study is that it will provide useful information to improve our understanding of insomnia and to enhance efficacy and efficiency of therapeutic approaches for a prevalent and costly health problem. The long-term objective is to contribute to the development and dissemination of evidence-based treatments for chronic insomnia and its common comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 years old or older
* Chronic insomnia(> 6 months)
* 3 nights or more per week with difficulties falling or staying asleep

Exclusion Criteria:

* Progressive or unstable medical condition directly interfering with sleep
* History of psychosis or bipolar disorder
* Alcohol/substance abuse within the past 12 months
* Use of medications interfering with sleep
* Presence of another sleep disorder (e.g., sleep apnea, restless legs syndrome/periodic limb movements)
* Irregular sleep-wake schedule

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2008-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Sleep/insomnia measures: sleep continuity (sleep latency, time awake after sleep onset, total sleep time); insomnia severity index; daytime functioning measures: fatigue, work/social adjustment, quality of life | pre, post, 6- and 12-month follow ups

SECONDARY OUTCOMES:
psychological/psychiatric measures: severity of anxiety (STAI) and depressive symptoms (BDI); mechanism/process measures | pre, post, 6- and 12-month follow ups

CONTACTS AND LOCATIONS:
Overall Officials: Charles M. Morin, PhD, Principal Investigator — Laval University
Locations (2):
- University of California at Berkeley, Berkeley, California, United States
- Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Sarfan LD, Morin CM, Harvey AG. Twelve-month follow-up: Comparative efficacy of cognitive therapy, behavior therapy, and cognitive behavior therapy for patients with insomnia. J Consult Clin Psychol. 2023 Oct;91(10):606-613. doi: 10.1037/ccp0000802. Epub 2023 Feb 23. PMID 36821333
- [Derived] Dong L, Soehner AM, Belanger L, Morin CM, Harvey AG. Treatment agreement, adherence, and outcome in cognitive behavioral treatments for insomnia. J Consult Clin Psychol. 2018 Mar;86(3):294-299. doi: 10.1037/ccp0000269. Epub 2017 Dec 21. PMID 29265834
- [Derived] Belanger L, Harvey AG, Fortier-Brochu E, Beaulieu-Bonneau S, Eidelman P, Talbot L, Ivers H, Hein K, Lamy M, Soehner AM, Merette C, Morin CM. Impact of comorbid anxiety and depressive disorders on treatment response to cognitive behavior therapy for insomnia. J Consult Clin Psychol. 2016 Aug;84(8):659-67. doi: 10.1037/ccp0000084. Epub 2016 Mar 10. PMID 26963600
- [Derived] Eidelman P, Talbot L, Ivers H, Belanger L, Morin CM, Harvey AG. Change in Dysfunctional Beliefs About Sleep in Behavior Therapy, Cognitive Therapy, and Cognitive-Behavioral Therapy for Insomnia. Behav Ther. 2016 Jan;47(1):102-15. doi: 10.1016/j.beth.2015.10.002. Epub 2015 Oct 19. PMID 26763501